CLINICAL TRIAL: NCT04335604
Title: An Open-label, Dose-finding, Phase I Study to Assess the Safety, Tolerability, and Pharmacokinetic-pharmacodynamic Profile of NOV140201 (JPI-547), a Dual Inhibitor of PARP/TNK in Patients With Advanced Solid Tumors
Brief Title: A Study of NOV140201 (JPI-547) in Subject With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Collaborators: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV140201-101
Record Dates: First submitted 2018-01-31; First posted 2020-04-06 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JPI-547 (Experimental)
  Interventions: Drug: JPI-547

INTERVENTIONS:
Drug: JPI-547 — The dose levels will be escalated following a 3+3 dose escalation scheme.

SUMMARY:
To assess the Safety, Tolerability, and Pharmacokinetic-pharmacodynamic Profile and efficacy of JPI-547 in patients with advanced solid tumor.

DETAILED DESCRIPTION:
This is an open-label, Phase 1 dose escalation and expansion study of NOV140201 (JPI-547) to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and the anti-tumor efficacy of JPI-547 in patients with advanced solid tumors after failure of standard of care.

Patients will be enrolled in two stages: a dose-escalation stage and an expansion phase. DLTs will be assessed as the primary endpoint in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 19 years old or above
* Patients that are histologically or cytologically confirmed advanced solid tumors and are refractory to or are able to receive standard of care
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy ≥12 weeks
* Individuals who volunteer to give to the written consent to the participation after listening to sufficient explanation for this clinical study

Exclusion Criteria:

* History of severe drug hypersensitivity or hypersensitivity to IP or similar class
* Patients who have the confirmed medical history or surgery/procedure history as the followings:

  1. History of major surgery requiring general anesthesia or assisted respiration within 4 weeks prior to baseline (within 2 weeks for video-assisted thoracoscopic surgery (VATS) or open-and-closed (ONC) surgery)
  2. Severe cardiovascular disease (eg. myocardial infarction or unstable angina pectoris) within 24 weeks prior to baseline
  3. New York Heart Association Class III or IV heart failure within 24 weeks prior to baseline
  4. Severe cerebrovascular disease within 24 weeks prior to baseline
  5. Pulmonary artery thrombosis, deep vein thrombosis, or clinically severe pulmonary disease within 24 weeks prior to baseline
  6. Infection requiring the administration of systemic antibiotics, antivirals or other uncontrolled Grade ≥3 Active infectious disease within 2 weeks prior to baseline
  7. Symptomatic interstitial lung disease
  8. Poor recovery from hematologic toxicities in previous anticancer treatment (eg. >4 weeks of Grade 3≥ toxicities)
  9. Individuals who receive bone marrow or stem cell transplant with a high dose of chemotherapy
* Individuals as accompanied by the following diseases:

  1. Hematologic malignancy other than lymphoma
  2. History of myelodysplastic syndrome (MDS) or pre-treatment cytogenetic test results indicative of the risk of MDS/acute myelocytic leukemia (AML)
  3. Patients with symptomatic with clinically significant or uncontrolled central nervous system (CNS) or brain metastasis (other than patients who discontinued the administration of systematic corticosteroid at least 4 weeks prior to baseline and who are radiologically and neurologically stable for ≥4 weeks)
  4. Patients with clinically significant abnormalities in the judgment of the investigator according to electrocardiogram findings
  5. Uncontrolled hypertension (systolic blood pressure>140mmHg or diastolic blood pressure >90mmHg)
  6. Bleeding diatheses
  7. History of active hepatitis B or C virus (hepatitis patients acceptable if HBV DNA and HCV RNA are <institutional lower limits)
  8. positive known human immunodeficiency virus (HIV)infection
  9. Severe neurological disorder and mental illness that may affect the study results in the opinion of the investigator
* Individuals who have the following medication history:

  1. Individuals with medication history of PARP inhibitors or TNK inhibitors (This applies only to Part 2.)
  2. Individuals receiving chemotherapy, biological therapy, retinoid therapy, immunotherapy, hormone therapy or therapeutic/palliative radiotherapy for the treatment of advanced solid tumors within 4 weeks prior to baseline (except for the individuals who received nitrosourea or mitomycin within 6 weeks prior to baseline and biological target antibody within 6 weeks prior to baseline)
  3. Patients requiring the continuous administration of non-steroidal anti-inflammatory drug (NSAID) with a high bleeding risk
  4. Patients requiring continuous administration of systemic corticosteroid equivalent to Prednisone >10 mg/day
  5. Individuals who received antithrombotics, including antiplatelets and anticoagulants within 2 weeks of baseline, or expecting to require the administration during the clinical study (the administration of low molecular weight heparin (LMWH) is allowed for the management and prevention of venous thrombosis during the clinical study.)
  6. Individuals who start the new administration or dose change of bisphosphonate within 30 days of baseline among patients with breast cancer and prostatic cancer in a dose expansion cohort within 30 days of baseline (bisphosphonate administered stably for 30 days before baseline is allowed.)
* Pregnant women, breastfeeding women, or female of childbearing potential and male who are not willing to practice abstinence or use appropriate contraception* during the clinical study and for 3 months after the administration of the IP
* Individuals who were administered other IPs or the investigational device within 4 weeks prior to baseline
* Individual considered ineligible or unavailable for this study for other reasons, in the opinion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) and Maximum tolerated dose (MTD) | 21days
  subjects will be treated and observed for DLT through the end of the first cycle

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of JPI-547 | 1 and 15 days
  to observe pharmacokinetic parameter
Peak Plasma Concentration (Cmax) of JPI-547 | 1 and 15 days
  to observe pharmacokinetic parameter
Time at maximum concentration(Tmax) of JPI-547 | 1 and 15 days
  to observe pharmacokinetic parameter
Half-life of JPI-547 | 1 and 15 days
  to observe pharmacokinetic parameter
Accumulation ratio of JPI-547 | 1 and 15 days
  to observe pharmacokinetic parameter

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University College of Medicine, Seoul